CLINICAL TRIAL: NCT00237159
Title: Effect of Zoledronic Acid in Patients With Prostate Cancer and Bone Metastasis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EDE07
Record Dates: First submitted 2005-10-09; First posted 2005-10-12 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Prostate Cancer Patients With Bone Metastasis
Keywords: Prostate cancer; Bone metastasis; Skeletal related event
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

ARMS (1):
- ZOL446 (Experimental)
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid
  Other Names: ZOL446

SUMMARY:
It is the aim of this clinical study to evaluate the skeletal-related event rate and tolerability of zoledronic acid in patients with prostate cancer patients and bone metastases.

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent
* A histologically confirmed diagnosis of carcinoma of the prostate
* Therapy with hormonal treatments (medical or surgical castration)
* Patients must have objective evidence of metastatic disease to bone.
* Adequate liver function - serum total bilirubin concentration less than 1.5 x upper limit of normal value
* ECOG performance status of 0, 1 or 2

Exclusion criteria:

* Bone pain which requires strong narcotic therapy with centrally acting analgesic agents.
* More than 3 bisphosphonate applications in patients history.
* Previous Radiation therapy to bone (including therapeutic radioisotopes such as strontium 89) within 3 months prior to Visit 2.
* Abnormal renal function as evidenced by

A calculated creatinine clearance < 30 ml/minute. Creatinine clearance (CrCl) is calculated using the Cockcroft-Gault formula:

CrCl= [140-age (years)] x weight (kg) {x 0.85 for female patients} [72 x serum creatinine (mg/dL)]

* Corrected (adjusted for serum albumin) serum calcium concentration < 8.0 mg/dl (2.00 mmol/L) or ≥ 12.0 mg/dl (3.00 mmol/L)
* Life expectancy < 6 months
* Patients with evidence in the six months prior to randomization of severe cardiovascular disease (defined as uncontrolled congestive heart failure), hypertension refractory to treatment, or symptomatic coronary artery disease uncontrolled by treatment
* Use of other investigational drugs (drugs not marketed for any indication) within 30 days prior to the date of randomization
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures.
* Recent (within 6 weeks) or planned dental or jaw surgery (e.g. extraction, implants)

Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2002-10; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Rate of skeletal complications | 3 months

SECONDARY OUTCOMES:
Time to first skeletal complication | 3 months
Bone pain | 3 months
Patients´ satisfaction with treatment | 3 months
Bone turnover parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals